CLINICAL TRIAL: NCT06150807
Title: Frequency and Risk Factors of Portal Vein Thrombosis in Neonate With Umbilical Catheter
Brief Title: Portal Vein Thrombosis in Neonate With Umbilical Catheter
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, esraa mostafa ahmed, MA Researcher, Assiut University
Other Study IDs: portal vein thrombosis
Record Dates: First submitted 2023-11-21; First posted 2023-11-29 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-11

CONDITIONS: Portal Vein Thrombosis
MeSH Terms: interventions — Ultrasonography, Doppler

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: ultrasound and doppler — Ultrasound examinations of the liver and spleen including color Doppler imaging of the portal veins, hepatic veins, splenic vein, and superior mesenteric vein will done in the Department of Pediatric

SUMMARY:
The aim of this study is to identify incidence of portal vein thrombosis after umbilical catheter and to identify the risk factor of this condition ,location of PVT and prognosis of PVT.

DETAILED DESCRIPTION:
The use of umbilical venous catheters (UVCs) in the neonatal period may be associated with severe complications including the occurrence of portal vein thrombosis (PVT )(1) The placement of an umbilical venous catheter (UVC) is a common procedure in neonatology and has multiple clinical indications driven by the need for quick and secure access for medication administration. Umbilical venous catheters allow quick access for administering drugs, blood products, fluids and parenteral nutrition to acutely ill neonates; however, they are have many complications. The most common complication is nosocomial sepsis ranging from 3% to 16%, followed by thromboembolism and catheter malposition in the heart, great vessels or portal system(2,3) The diagnosis is made by abdominal Doppler ultrasonography . In the cases with portal venous thrombosis, the location, extent, and size of the thrombus were recorded occlusive was defined by hyperechogenic thrombus replacing the entire lumen and no-flow in color Doppler or Partial which defined by non-occlusive hyperechogenic intraluminal thrombus and persistent stream in color Doppler.(4) A prospective observational study of newborns, who were admitted to the Neonatal intensive care Unit Assiut University Children's Hospital ,neonates who had undergo UVC for any cause between 10/2023 to 9/2024 will enroll in these study with serial ultrasonography of the UVC to determine the incidence and location of thrombi in infants after umbilical catheterization.

All cases included in the study will be evaluated by Birth weight, gender, gestational age, type of catheter, duration of catheter use, types of infused fluids, and location of the catheter tips (UVC), Ultrasound examinations of the liver and spleen including color Doppler imaging of the portal veins, hepatic veins, splenic vein, and superior mesenteric vein will done in the Department of Pediatric Diagnostic Imaging by a radiologist after removal of the catheter and in case of PVT subsequent serial U/S will preformed until clot resolution.

ELIGIBILITY:
Inclusion Criteria:

* the study population: all neonates with UVC, who will admitted to the Neonatal intensive care Unit Assiut University Children's Hospital had undergo UVC for any cause between 10/2023 to 9/2024 limited to diagnosis established in neonates <28-day chronological age.

Exclusion Criteria:

* Neonate who has PVT but not had UVC before .

Ages: 1 Day to 28 Days | Sex: All
Age Groups: Child
Study Population: all neonates with UVC, who will admitted to the Neonatal intensive care Unit Assiut University Children's Hospital had undergo UVC for any cause between 10/2023 to 9/2024 limited to diagnosis established in neonates <28-day chronological age.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2023-12-20 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
Frequency and risk factors of portal vein thrombosis in neonate with umbilical catheter | baseline
  Identify incidence of portal vein thrombosis after umbilical catheter,Identify the risk factor of this condition ,location of PVT and prognosis of PVT.

REFERENCES:
- [Background] Salimi M. Comparison of beta-adrenoceptor blocking properties of sotalol, oxprenolol, propranolol and pindolol on rabbit intestinal smooth muscle. Pharmacology. 1975;13(5):441-7. doi: 10.1159/000136936. PMID 1802